CLINICAL TRIAL: NCT02764983
Title: Efficacy of a Driving Program on Safe Community Mobility for Combat Veterans
Brief Title: Occupational Therapy Driving Intervention for Returning Combat Veterans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 652-2011; IRB201702264 (Other: University of Florida); JW140063 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2016-04-18; First posted 2016-05-06 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Traumatic Brain Injury (TBI); Post Traumatic Stress Disorder (PTSD)
Keywords: Combat Veterans; Automobile Driving; Fitness to Drive
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Group (Active Comparator): Participants in this group will have the following performed: Institute of Mobility Activity and Participation (I-MAP's) clinical battery of tests and a simulated driving test, a Brief Driving Behavior Interview, Propensity for Angry Driving Scale, Clinical Driving Assessment, Community Integration Questionnaire, and a Satisfaction with Life Questionnaire. Driving safety professional, three x 1 hour sessions to discuss traffic safety, rules of the road, defensive driving, driving under influence, driver attitudes and safety. Additionally, the study will obtain real world driving data from the Department of Motor Vehicles (public records) which will include citations, violations, and recorded collisions/ crashes.
  Interventions: Behavioral: Driving Behavior Interview; Behavioral: Fitness-to-Drive Screening Measure; Other: Clinical Driving Assessment; Behavioral: Propensity for Angry Driving Scale; Behavioral: Community Integration Questionnaire; Behavioral: Satisfaction with Life Questionnaire; Procedure: Driving simulator evaluation
- Experimental Group (Experimental): Participants in this group will have the following performed: Institute of Mobility Activity and Participation (I-MAP's) clinical battery of tests and a simulated driving test, a Brief Driving Behavior Interview, Propensity for Angry Driving Scale, Clinical Driving Assessment, Community Integration Questionnaire, and a Satisfaction with Life Questionnaire. Occupational Therapy Driving Intervention (OT-DI) consisting of three x 1 hour sessions to review explicit driving errors, strategies to mitigate errors, and driving simulator with feedback. The study will also obtain real world driving data from the Department of Motor Vehicles (public records) which includes citations, violations, and recorded collisions/crashes.
  Interventions: Behavioral: Driving Behavior Interview; Behavioral: Fitness-to-Drive Screening Measure; Other: Clinical Driving Assessment; Behavioral: Propensity for Angry Driving Scale; Behavioral: Community Integration Questionnaire; Behavioral: Satisfaction with Life Questionnaire; Procedure: Driving simulator evaluation
- Caregiver Control Group (Active Comparator): Participants in this group will perform the following: Fitness-to-Drive Screening Measure(FTDS) will be filled out at baseline and again at the end of the study.
  Interventions: Behavioral: Fitness-to-Drive Screening Measure
- Caregiver Experimental Group (Active Comparator): Participants in this group will perform the following: Fitness-to-Drive Screening Measure(FTDS) will be filled out at baseline and again at the end of the study.
  Interventions: Behavioral: Fitness-to-Drive Screening Measure
- Focus Group Discussion Interview Guide (Other): This group will comprise of a subset of the control and experimental groups. A focus group with 8 participants (4 with Traumatic Brain Injury/Post Traumatic Stress Disorder and 4 with orthopedic conditions). The focus group will meet once for a discussion which will be guided with a semi-structured interview that will explore the driving behavior prior to war, during war and post-deployment. Responses will be outlined in an intervention matrix.
  Interventions: Other: Focus Group Discussion Interview Guide

INTERVENTIONS:
Behavioral: Driving Behavior Interview — This will be completed thrice, at baseline, post-test1 and at post-test2
  Arms: Control Group; Experimental Group
Behavioral: Fitness-to-Drive Screening Measure — This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test1)
  Arms: Caregiver Control Group; Caregiver Experimental Group; Control Group; Experimental Group
Other: Clinical Driving Assessment — Clinical Driving Assessment includes Optec vision screening, Useful Field of View, Range of Motion, Strength. This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test1)
  Arms: Control Group; Experimental Group
Behavioral: Propensity for Angry Driving Scale — This questionnaire will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test1)
  Other Names: Road rage questionnaire
  Arms: Control Group; Experimental Group
Behavioral: Community Integration Questionnaire — This questionnaire will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test1)
  Arms: Control Group; Experimental Group
Behavioral: Satisfaction with Life Questionnaire — This questionnaire will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test1)
  Arms: Control Group; Experimental Group
Procedure: Driving simulator evaluation — The driving simulator evaluation uses a driving simulator with simulated drives engineered to address Veteran driving concerns such as reactions to other drivers and road conditions (e.g., debris). The simulator is used at baseline and post-tests 1 and 2. The intervention sessions (X3) also occur using simulator.
  Arms: Control Group; Experimental Group
Other: Focus Group Discussion Interview Guide — Focus group discussion will occur once using the interview guide
  Arms: Focus Group Discussion Interview Guide

SUMMARY:
Driving is a portal into general life functioning, and impaired driving skill can pose a serious threat to the combat veterans (CV), passengers and others; and involves increased risk of subsequent injuries, medical expenses and legal sequelae. Motor vehicle crashes (MVC) among post deployed CV are one of the top four causes of injury and disability, hospitalization, and outpatient visits across the military, and are a leading cause of death among Army service members. The risk of motor vehicle (MV) death is significantly increased in years immediately following return from the battlefield. In sum, the effects of Traumatic Brain Injury (TBI)/ Post Traumatic Stress Disorder (PTSD) and other blast related injuries, combined with the "battlefield" mindset and lack of community reintegration programs place CV at risk for MVC and fatalities. On-road assessments, the gold standard, presents a risk for crash or adverse advents in this population of CV. Alternately, simulated driving evaluation measures driving performance in a safe, accurate and objective manner with evidence of absolute and relative validity when compared to real world (on-road) driving. Knowing participants can or cannot safely resume driving, and providing rehabilitation for those with a potential for resuming safe driving could result in: increased safe driving behaviors; avoidance of injuries, collisions, citations and participants residua; and resuming safe driving with its attendant benefits in the realms of family functioning, participation in society and satisfaction with life. The overarching objective of this proposal is to discern, after clinical and simulated driving performance testing , if Occupational Therapy Driving Intervention (OT-DI) can improve the safe driving performance (less errors) over the short term (immediately following intervention) and intermediate term (3 months).

DETAILED DESCRIPTION:
This research study is being done to determine if Occupational Therapy Driving Intervention (OT-DI) can improve the safe driving performance (less errors) over the short term (immediately following intervention) and intermediate term (3 months).

Baseline testing-Pre-test 1-- will include clinical battery of tests and a simulated driving test, a Brief Driving Questionnaire, Community Integration Questionnaire, and a Satisfaction with Life Questionnaire. Caregivers/ family members will rate the participants' driving behaviors using a Fitness-to-Drive Screening Measure( FTDS). After baseline testing the 60 participants (and 60 associated caregivers) will be randomly assigned to a balanced intervention group (15 participants with Traumatic Brain Injury (TBI)/ Post Traumatic Stress Disorder (PTSD) and 15 participants with orthopedic conditions and caregivers) and a control group (15 with TBI/PTSD and 15 with orthopedic conditions and caregivers).

The intervention group receives Occupational Therapy Driving Intervention (OT-DI), consisting of three x 1 hour sessions will include: Session 1: Driving evaluator reviews explicit driving errors with participants; Session 2: Driving evaluator provide tailored strategies to mitigate errors; Session 3: Participants drive simulator with targeted feedback from driving evaluator.

The control group will receive, from a driving safety professional, three x 1 hour general safety sessions (Session 1: General traffic safety discussion; Session 2: Rules of the road and knowledge of the road discussion; Session 3: drive the simulator without any feedback from traffic safety professional). Immediately after session 3, Post-test 1 will occur using the same standardized protocol outlined for baseline testing. Post-test 2 will consist of testing with the same standardized protocol as administered during baseline testing. Caregivers/ family members will rate the participant driving behaviors using the FTDS. In addition, the investigators will obtain driving data from the Department of Motor Vehicles which will include: citations, violations, driving mishaps, and crashes that have occurred for each participant.

ELIGIBILITY:
Inclusion Criteria:

* A combat veteran with polytrauma (mild traumatic brain injury/with an accompanying post traumatic stress disorder (PTSD), traumatic limb amputation/ fractures), who drove prior to the injury/condition;
* have a valid driver's license or are eligible for a driver's license;
* are community dwelling;
* may experience self, physician or other clinical staff identified issues with driving behaviors;
* have a history of citations, violations or other driving mishaps in real world driving;
* have potential for following driving safety recommendations (Mini Mental State Examination, (MMSE 24/30);
* have potential for following community integration strategies (MMSE 24/30);
* are able to participate in driving evaluation battery.

Exclusion Criteria:

* A combat veteran diagnosed with a severe psychiatric (psychoses) or physical conditions (missing both arms and/or legs) that will limit ability to drive;
* have multiple psychotropic medications that may impact mental or physical (due to side-effects) functioning as per the consulting physician;
* have severe, irremediable medical conditions (severe TBI) as per the consulting physician;
* pregnant females (as determined by a urine test) or those planning pregnancy;
* VA Employees; and
* veterans who have received rehabilitation services for TBI/PTSD and who show, as per the screening of the driving rehabilitation specialist, a poor prognosis for improvement based on a driving intervention.

Inclusion Criteria for Caregivers:

* ability to complete a driving questionnaire pre and post intervention.

Exclusion Criteria for Caregivers:

* the presence of a cognitive or physical impairment that would hinder participants ability to complete the questionnaires or make an active contribution.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Driving errors changes between the groups at baseline, months 2 and 3 | Changes in baseline months 2 and 3
  Determine if the Occupational Therapy Driving Intervention (OT-DI) reduces driving errors in the intervention group.

SECONDARY OUTCOMES:
Perceptions of Combat Veterans regarding driving performance | Occurs approximately 2 months after baseline (75 minutes)
  Semi-structured interview questions will be used to guide the focus group discussions. The results will be outlined in an intervention matrix which will be used to address specific driving errors and the behavior underlying those errors in the intervention process.
Change in driving records from baseline and at 11months | From baseline (approximately 11months)
  Driving records from the Department of Motor Vehicle will be collected to determine if driving errors have reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Winter, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Classen S, Winter S, Monahan M, Yarney A, Link Lutz A, Platek K, Levy C. Driving Intervention for Returning Combat Veterans. OTJR (Thorofare N J). 2017 Apr;37(2):62-71. doi: 10.1177/1539449216675582. Epub 2016 Nov 29. PMID 27830643